CLINICAL TRIAL: NCT00470639
Title: A Comparison of Left vs. Right Prefrontal Cortex Transcranial Magnetic Stimulation as a Treatment for Bipolar Depression
Brief Title: Transcranial Magnetic Stimulation for Bipolar Depression
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07103
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Bipolar Depression
Keywords: TMS; Treatment; Bipolar; Efficacy
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMS (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham (Sham Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation

SUMMARY:
This is a study to assess the effectiveness of repetitive transcranial magnetic stimulation (rTMS) as a treatment for depressed adults with bipolar disorder.

In rTMS high-intensity, fluctuating magnetic fields non-invasively stimulate the cortex of the brain depolarising neurons. No anaesthetic is required and the treatment in subconvulsive. Recent studies suggest that rTMS can be an effective treatment for depressive illness in adults (Loo and Mitchell et al, 2005) and appears to be quite safe.

Most of the published studies to date have focused on unipolar depression. There is limited data of TMS use in bipolar depression. Eg. Pilot study by Nahas Z, Kozel FA, Li X, Anderson B, George MS.in 2003, which was negative.

The investigators wish to assess this in a sham-controlled study of adults. The investigators hypothesise that both left and right sided rTMS will have an antidepressant effect superior to sham in this population.

DETAILED DESCRIPTION:
Inpatients and outpatients with major depressive episodes as part of either bipolar I or II illness will be eligible. In the event that patients (in any arm) have no significant response after a defined period, they will shift to an open phase where they will receive left prefrontal 10Hz stimulation. Thus all participants will have the opportunity to receive active treatment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Major Depressive Episode of no more than 3 years.
* Diagnosis of bipolar I or II disorder
* Montgomery-Asberg Depression Rating Scale score of 20 or more.
* Aged over 18
* May or may not be taking antidepressant medication.

Exclusion Criteria:

* Patient not able to give informed consent.
* Failure to respond to ECT in current episode of depression.
* Significant other Axis I psychiatric disorders e.g. schizophrenia.
* In imminent physical or psychological danger, or needs rapid clinical response due to inanition, psychosis or high suicide risk.
* Comorbid substance abuse or dependence
* History of neurological illness e.g. epilepsy; neurosurgical procedure
* Metal in the cranium, a pacemaker, cochlear implant, medication pump or other electronic device.
* Women of child-bearing age in whom pregnancy cannot be ruled out.
* Patients with a history of mood 'switching' in response to other treatments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
All measures at baseline and at the end of each week of treatment in the blind phase and after every 2 weeks of treatment in the open phase. | weekly
Montgomery-Asberg Depression Rating Scale (MADRS) | Weekly
Clinical Global Impressions Scale (CGI) | Weekly

SECONDARY OUTCOMES:
Patient Global Improvement scale | Weekly
Young Mania Rating Scale | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, FRANZCP, MD, Principal Investigator — University of New South Wales; William Lyndon, FRANZCP, Study Director — University of Sydney
Locations (2):
- Australia (2):
  - Black Dog Research Institute, Sydney, New South Wales
  - Northside Clinic, Sydney, New South Wales

REFERENCES:
- [Background] Nahas Z, Kozel FA, Li X, Anderson B, George MS. Left prefrontal transcranial magnetic stimulation (TMS) treatment of depression in bipolar affective disorder: a pilot study of acute safety and efficacy. Bipolar Disord. 2003 Feb;5(1):40-7. doi: 10.1034/j.1399-5618.2003.00011.x. PMID 12656937
- [Background] Loo CK, Mitchell PB. A review of the efficacy of transcranial magnetic stimulation (TMS) treatment for depression, and current and future strategies to optimize efficacy. J Affect Disord. 2005 Nov;88(3):255-67. doi: 10.1016/j.jad.2005.08.001. Epub 2005 Sep 2. PMID 16139895